CLINICAL TRIAL: NCT05554250
Title: Turkish Validity and Reliability Study of Reward-Based Eating Drive (RED) Scale
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, CANAN ALTINSOY, Araştırma Görevlisi, Hacettepe University
Other Study IDs: RecepTayyipErdoganU
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Eating Disorders; Eating Habit; Obesity
Keywords: validity; measuring tool; reliability; obesity; eating disorder; eating habits; reward
MeSH Terms: conditions — Feeding and Eating Disorders; Feeding Behavior; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obese patients: The population of the study consisted of individuals who applied to the Diet Polyclinic of a hospital, and the sample consisted of 500 individuals who applied to the Diet Polyclinic and met the research criteria.

SUMMARY:
This research; The Turkish validity and reliability study of the "Reward-Based Eating Impulse Scale-13" developed by Ashley E. Mason was conducted to provide a new measurement tool for our country. At the same time, the study will provide a database for intervention studies to eliminate the effects of reward-based eating urge. Identifying reward-based eating in the middle and lower ranges of the eating disorder spectrum may contribute to halting the growing obesity epidemic. The Reward-Based Eating Impulse Scale will help researchers and clinicians to identify individuals who lack control over eating, cannot feel full, and are constantly preoccupied with eating.

DETAILED DESCRIPTION:
Today, with the spread of Western-style nutrition, pleasure-based nutrition is increasing. Especially the easy access to delicious foods with high sugar, fat and salt content encourages individuals to have a diet based on pleasure rather than energy needs (Lowe, 2003). Reward-based eating behavior can occur in order to reinforce and strengthen positive emotions such as happiness and joy, or to suppress negative emotions such as stress and anxiety (Evers et al., 2013). If reward-based eating is repeated frequently in response to positive or negative emotions, it may underlie the development of eating pathology and binge eating disorder. Therefore, researchers working in the context of health behaviors, nutrition, and metabolic health triad evaluate reward-based eating before, during, and after interventions targeting changes in health behavior (Forman et al., 2013; Mason et al., 2016; Stevenson et al., 2018).

Individuals' degree of reward-based eating is measured by evaluating behaviors such as uncontrolled eating, food craving, food addiction, restrictive eating, and binge eating. Each of the scales focuses on a different aspect of problematic eating behavior (Price et al., 2015; Vainik et al., 2015). For example, the Yale Scale of Eating Addiction considers eating behavior in terms of the Diagnostic and Statistical Manual of Mental Disorders (DSM) criteria. Therefore, only when the problem becomes pathological can they evaluate reward-based eating. Similarly, the Binge Eating Scale evaluates when problematic eating behavior is severe. The Nutrient Power Scale and the Tasty Eating Motivation Scale, on the other hand, evaluate the causes of binge eating behavior and food choice in the environmental context and focus on a less problematic process than the others (Burgess et al., 2014; Davis, 2013; Gearhardt, 2016; Lowe et al., 2009) . Each developed scale better measures one aspect of reward-based eating behavior. For example, a scale that assesses the urge to eat may measure less uncontrolled eating. While the Dutch Eating Behavior Questionnaire measures emotional eating better, it measures less uncontrolled eating and binge eating (Gormally et al., 1982). All sub-dimensions indicate the stages of the person's pathology of binge eating. For example, people with high impulsivity about eating use food to cope with emotions over time and eventually develop binge eating disorder. Theoretical and experimental evidence suggests that none of these scales comprehensively assess reward-based eating (Davis, 2013).

In order to comprehensively evaluate this issue, the Reward-Based Eating Impulse Scale (RED-9) was developed by Epel et al., which aims to address all spectrums of reward-based eating (Epel et al., 2014). RED-9 is associated with body mass index (BMI) and also predicts changes in BMI over time. In a study of obese women, food craving was shown to be associated with higher RED-9 scores. Although RED-9 is short and simple to apply, it is unclear whether it assesses the full spectrum of reward-based eating (Mason et al., 2015; Mason et al., 2016). RED-13 assesses three dimensions of reward-based eating: lack of control over eating, inability to achieve satiety, and constant preoccupation with food. It has been shown that reduction in reward-based eating behavior may mediate the effect of obesity treatment on weight loss.

This research; The Turkish validity and reliability study of the "Reward-Based Eating Impulse Scale-13" developed by Ashley E. Mason was conducted to provide a new measurement tool for our country. At the same time, the study will provide a database for intervention studies to eliminate the effects of reward-based eating urge. Identifying reward-based eating in the middle and lower ranges of the eating disorder spectrum may contribute to halting the growing obesity epidemic. The Reward-Based Eating Impulse Scale will help researchers and clinicians to identify individuals who lack control over eating, cannot feel full, and are constantly preoccupied with eating.

Research Question Is the "Reward-based Eating Drive Scale (RED)" a valid and reliable measurement tool for Turkish society?

ELIGIBILITY:
Inclusion Criteria:

* Persons who are at least 18 years old, have a body mass index of 30 kg/m2 and above, are at least primary school graduates, can communicate verbally and agree to participate in the research.

Exclusion Criteria:

* Persons with psychiatric illness who could not communicate, who could not read and understand Turkish, and who did not have the skills to read and understand the questionnaire were excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Obese patients
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-12-28 (Estimated)

PRIMARY OUTCOMES:
Reward-based Eating Scale | 30 minutes
  The data of the research are obtained by "Personal Information Form" and "Reward-based Eating Drive Scale (RED-13)". High scores from the scale will help determine the risk group.

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdogan University, Rize, İslampasa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No